CLINICAL TRIAL: NCT07265466
Title: A Phase 1 Clinical Trial to Evaluate the Safety and the Pharmacokinetic and Pharmacodynamic Interactions Between JP-1366 and Clopidogrel, Aspirin, Atorvastatin and Apixaban in Healthy Volunteers.
Brief Title: to Evaluate the Safety and the Pharmacokinetic and Pharmacodynamic Interactions Between JP-1366 and Clopidogrel, Aspirin, Atorvastatin and Apixaban
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-106
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Drug Drug Interaction (DDI)
MeSH Terms: interventions — Clopidogrel; Aspirin; Atorvastatin; apixaban

STUDY DESIGN:
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): JP-1366 and clopidogrel
  Interventions: Drug: JP-1366 and clopidogrel
- Part 2 (Experimental): JP-1366 and aspirin
  Interventions: Drug: JP-1366 and aspirin
- Part 3 (Experimental): JP-1366 and atorvastatin
  Interventions: Drug: JP-1366 and atorvastatin
- Part 4 (Experimental): JP-1366 and apixaban
  Interventions: Drug: JP-1366 and apixaban

INTERVENTIONS:
Drug: JP-1366 and clopidogrel — A randomized, open label, multiple-dosing, 6-sequence, 3-period, 3-treatment, crossover design
  Arms: Part 1
Drug: JP-1366 and aspirin — An open-label, multiple-dosing, fixed sequence, 3-period design
  Arms: Part 2
Drug: JP-1366 and atorvastatin — An open-label, multiple-dosing, fixed sequence, 3-period design Period 1: Atorvastatin
  Arms: Part 3
Drug: JP-1366 and apixaban — An open-label, multiple-dosing, fixed sequence, 3-period design
  Arms: Part 4

SUMMARY:
to Evaluate the Safety and the Pharmacokinetic and Pharmacodynamic Interactions between JP-1366 and Clopidogrel, Aspirin, Atorvastatin and Apixaban

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged ≥ 19 years to < 65 years at the time of screening
* Subjects who weigh ≥ 50 kg (or ≥ 45 kg in the case of females) with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2
* Subjects who have voluntarily decided to participate after fully understanding the clinical trial based on the detailed explanation given, and have provided written informed consent before the screening procedure.

Exclusion Criteria:

* Subject who has a clinically significant history of disease in the liver, kidneys, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hematopoietic and oncological system, or cardiovascular system.
* The Subject who has a clinically significant bleeding or a history of congenital or acquired bleeding disorders such as hemophilia
* Subject who has a history of gastrointestinal disorders (e.g., Crohn's disease, ulcerative disease, etc.) or surgery (excluding appendectomy, hernia repair, endoscopic polypectomy, or hemorrhoidectomy, fissure, or fistula surgery) that may affect the absorption of the investigational product.
* The subject who has a hereditary disorder (galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption etc.).
* Screening laboratory test showing any of the following abnormal laboratory results
* Subjects who are judged unsuitable to participate in the study in the opinion of the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
[Part 1] Change in P2Y12 Reaction Unit (PRU) from baseline on day 8 | baseline on day 8
  Change in P2Y12 Reaction Unit (PRU)
[Part 2] Emax of arachidonic acid-induced platelet aggregation | up to 48 hours post-dose on Day 1
  Emax of arachidonic acid-induced platelet aggregation
[Part 2] AUEC0-24 of arachidonic acid-induced platelet aggregation | up to 48 hours post-dose on Day 1
  AUEC0-24 of arachidonic acid-induced platelet aggregation
[Part 2] Cmax,ss of JP-1366 | up to 24 hours post-dose on Day 5
  Cmax,ss of JP-1366
[Part 2] AUCτ,ss of JP-1366 | up to 24 hours post-dose on Day 5
  AUCτ,ss of JP-1366
[Part 2] Cmax of Aspirin | up to 48 hours post-dose on Day 1
  Cmax of Aspirin
[Part 2] AUClast of Aspirin | up to 48 hours post-dose on Day 1
  AUClast of Aspirin
[Part 3] Cmax,ss of JP-1366 | up to 24 hours post-dose on Day 5
  Cmax,ss of JP-1366
[Part 3] AUCτ,ss of JP-1366 | up to 24 hours post-dose on Day 5
  AUCτ,ss of JP-1366
[Part 3] Cmax,ss of Atorvastatin | up to 24 hours post-dose on Day 5
  Cmax,ss of Atorvastatin
[Part 3] AUCτ,ss of Atorvastatin | up to 24 hours post-dose on Day 5
  AUCτ,ss of Atorvastatin
[Part 4] Emax of Anti-Factor Xa activity | up to 48 hours post-dose on Day 5
  Emax of Anti-Factor Xa activity
[Part 4] AUEC0-12 of Anti-Factor Xa activity | up to 48 hours post-dose on Day 5
  AUEC0-12 of Anti-Factor Xa activity
[Part 4] Cmax,ss of JP-1366 | up to 24 hours post-dose on Day 5
  Cmax,ss of JP-1366
[Part 4] AUCτ,ss of JP-1366 | up to 24 hours post-dose on Day 5
  AUCτ,ss of JP-1366
[Part 4] Cmax,ss of Apixaban | up to 12 hours post-dose on Day 5
  Cmax,ss of Apixaban
[Part 4] AUCτ,ss of Apixaban | up to 12 hours post-dose on Day 5
  AUCτ,ss of Apixaban

CONTACTS AND LOCATIONS:
Locations (1):
- Cha University Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No